CLINICAL TRIAL: NCT06205966
Title: A Randomized, Double Blind, Placebo-controlled Study to Investigate the Effect of Probiotics (L. Reuteri ATCC PTA 5289 and L. Reuteri DSM 17938) on Symptoms of Viral Upper Respiratory Tract Infections in Children
Brief Title: A Study to Investigate the Effect of Probiotics (L. Reuteri ATCC PTA 5289 and L. Reuteri DSM 17938) on Symptoms of Viral Upper Respiratory Tract Infections in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Milosevits Gergely (Other)
Responsible Party: Sponsor-Investigator, Milosevits Gergely, Principal Investigator, Szent Miklós Szolgálat Kft.
Organization: Szent Miklós Szolgálat Kft. (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SzentMiklósSzolgálatKft.
Record Dates: First submitted 2024-01-02; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Virus Diseases in Children

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Active Comparator): Study product containing L. reuteri (PTA5289 and DSM 17938) taken orally once in the morning and once in the evening, each time 5 drops.
  Interventions: Dietary Supplement: BioGaia Pharax (L. reuteri PTA 5289 and DSM 17938)
- Placebo (Placebo Comparator): Placebo taken orally once in the morning and once in the evening, each time 5 drops.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: BioGaia Pharax (L. reuteri PTA 5289 and DSM 17938) — BioGaia Pharax drops (with PTA5289 and DSM 17938) with vitamin D3 will be manufactured and delivered by BioGaia AB as oil suspension.
  Arms: Probiotics
Other: Placebo — Placebo product contains vitamin D3 and is identical to the active product but lacks L. reuteri.
  Arms: Placebo

SUMMARY:
This study investigates the effect of Lactobacillus reuteri probiotic strains (ATCC PTA 5289 and DSM 17938) on symptoms of viral upper-respiratory tract infections in children.

DETAILED DESCRIPTION:
Lactobacillus reuteri probiotic strains (ATCC PTA 5289 and DSM 17938) have been shown to significantly reduce the number of febrile days and pain severity in upper respiratory tract infections in children aged six months to 5 years. The investigator's planned study complements this earlier publication by significantly increasing the number of cases and expanding the age range studied including children from 4 to 17 years of age diagnosed with viral upper respiratory-tract infection.

ELIGIBILITY:
Inclusion Criteria:

* Children with symptoms of upper respiratory tract infection (coughing/fever/sneezing/runny or congested nose/pharynx pain)
* Any gender
* Age from 4 years to 17 years
* Signing a informed consent form by at least one parent, foster parent or guardian after patient information and by children aged over 6 years
* Negative Strep test

Exclusion Criteria:

* Use of antibiotics or probiotics in the 10 days prior to study enrolment
* Use of a probiotic other than the test sample during the study
* Eight or more otitis media within 12 months
* Two or more bacterial sinusitis within 12 months
* Two or more pneumonia episodes within 12 months
* History of two or more invasive infections (meningitis, cellulitis, osteomyelitis, septicaemia)
* Chronic diarrhea
* Recurrent deep skin or organ abscesses
* Persistent superficial candidiasis
* Use of antibiotics for two months or more to treat respiratory infections within 12 months
* Gastroesophageal reflux
* Perennial (e.g., dust mite or mold) or current seasonal hay fever allergy
* Primary or secondary ciliary dyskinesia
* Congenital malformations of the respiratory tract

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 142 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Time to healing, defined as number of hours until absence of symptoms (fever, runny nose, stuffy nose, sneezing, sore throat, cough, feeling tired) as well as absence of use of Non-steroidal anti-inflammatory drugs (NSAIDs) | 10 days

SECONDARY OUTCOMES:
Duration of symptoms (runny nose, stuffy nose, sneezing, sore throat, cough, feeling tired) | 10 days
Severity of symptoms (runny nose, stuffy nose, sneezing, sore throat, cough, feeling tired) recorded in a "Symptom Diary". | 10 days
  On a scale from 1 to 8.
Duration of fever, defined as the total number of hours that the child has a core temperature >38oC measured twice per day. | 10 days
Amount of NSAIDs used. | 10 days
Number of children receiving antibiotic treatment in each treatment group. | 10 days
Total amount of days of antibiotic use during the study, reported during the whole duration of the study in a the "Symptom Diary". | 10 days
Number of unplanned medical visits (other than "Visit 1 and 2"). | 10 days
  This outcome is defined as the total amount of medical office visits or emergency visits.
Days of absences from day care center/school. | 10 days
  This outcome is defined as the total amount of days of absences from the day care centre during the study, due to the presence of episodes of URTI.

CONTACTS AND LOCATIONS:
Locations (1):
- Szent Miklós Szolgálat Kft., Szigetszentmiklós, Pest County, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maya-Barrios A, Lira-Hernandez K, Jimenez-Escobar I, Hernandez L, Ortiz-Hernandez A, Jimenez-Gutierrez C, Lopez-Velazquez G, Gutierrez-Castrellon P. Limosilactobacillus reuteri ATCC PTA 5289 and DSM 17938 as adjuvants to improve evolution of pharyngitis/tonsillitis in children: randomised controlled trial. Benef Microbes. 2021 Apr 12;12(2):137-145. doi: 10.3920/BM2020.0171. Epub 2021 Apr 1. PMID 33789556